CLINICAL TRIAL: NCT06185218
Title: The Effect of Different Injection Site Maps on Intravesical Botulinum Toxin of Bladder
Brief Title: Different Injection Site Maps & Intravesical Botulinum Toxin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAEK/08.11.2023.530
Record Dates: First submitted 2023-11-28; First posted 2023-12-29 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-02

CONDITIONS: Bladder Disease
Keywords: Botulinum Toxin; overactive bladder; interstitial cystitis
MeSH Terms: conditions — Urinary Bladder Diseases; Urinary Bladder, Overactive; Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAP 1 (Posterior wall only) (Active Comparator): Type 1 map injection will be used to bladder in one session. In this arm, Botulinum toxin type A injection will be apply to non-trigonal only posterior wall of bladder. The application will be done with cystoscopy and, 20 different point will be aimed. Totally 100 IU Botulinum toxin type A will be applied.
  Interventions: Other: Intravesical Botulinum Toxin
- MAP 2 (Posterior wall + bilateral side walls) (Active Comparator): Type 2 map injection will be used to bladder in one session. In this arm, Botulinum toxin type A injection will be apply to non-trigonal posterior wall + bilateral side walls of bladder. The application will be done with cystoscopy and, 20 different point will be aimed. Totally 100 IU Botulinum toxin type A will be applied.
  Interventions: Other: Intravesical Botulinum Toxin
- MAP 3 (Non-trigonal all walls) (Active Comparator): Type 3 map injection will be used to bladder in one session In this arm, Botulinum toxin type A injection will be apply to non-trigonal all walls of bladder. The application will be done with cystoscopy and, 20 different point will be aimed. Totally 100 IU Botulinum toxin type A will be applied.
  Interventions: Other: Intravesical Botulinum Toxin

INTERVENTIONS:
Other: Intravesical Botulinum Toxin — Botulinum Toxin injections will be made into the bladder.

SUMMARY:
Botulinum toxin injection into the bladder is used in current practice in urological diseases such as overactive bladder or interstitial cystitis. As far as is known, botulinum toxin injection sites have not been clearly defined. In this study, investigators are planning to compare botulinum toxin effectiveness with different injection site maps.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Interstitial cystitis patients
* Overactive bladder

Exclusion Criteria:

* younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Overactive bladder-V8 questionnaire will be used for efficacy of treatment. | Estimated 1 month for every patient after treatment.
  The questionnaire contains 8 questions and every question may be scored between 0 and 5. Additionally, male gender get 2 points more. Therefore, a patient may be get between 0 and 42 points. More score means worse complaint.
Urodynamics test will be assessed for efficacy of treatment. | Estimated 1 month for every patient after treatment.
  Possible bladder contractions and residual volume will be measured in urodynamic testing to demonstrate effectiveness after treatment. The lack of pathological bladder contractions and normal residual urine mean better for patient and, show improving.

IPD SHARING:
Plan to Share IPD: Undecided